CLINICAL TRIAL: NCT00209430
Title: GEHC Has Decided Not to Provide This Detail But Will Rely on the Brief Title.
Brief Title: Renal Effects of Two Iodinated Contrast Media in Patients at Risk Undergoing Coronary Angiography
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: DXV405
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2007-10

CONDITIONS: Coronary Artery Disease; Renal Impairment
Keywords: Iodixanol; Iopamidol; coronary angiography; Contrast media-induced nephropathy
MeSH Terms: conditions — Coronary Artery Disease; Renal Insufficiency

INTERVENTIONS:
Drug: Iodixanol 320 mgI/mL

SUMMARY:
The main purpose of this study is to evaluate and compare the effects on kidney function of two contrast media, the iso-osmolar iodixanol and the low-osmolar iopamidol in patients at risk of kidney damage associated with the injection of contrast media. A standard hydration procedure, based on available guidelines will be given to all patients to prevent negative effects on the kidneys. Serum creatinine (SCr ) concentrations will be measured before and up to 7 days after contrast media administration to evaluate the effects on renal function.

DETAILED DESCRIPTION:
GEHC has decided not to provide this detail

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a combination of diabetes mellitus (type I or II) and renal impairment, defined as serum creatinine (SCr ) ≥150 µmol/L (1.7 mg/dL) for men and ≥133 µmol/L (1.5 mg/dL) for women or creatinine clearance (CrCl) ≤ 50 mL/min calculated according to Cockroft-Gault formula, referred for coronary angiography with or without PCI.

Exclusion Criteria:

* Concurrent administration of potentially nephroprotective or nephrotoxic drugs is not allowed. Subjects undergoing dialysis or kidney transplant will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408
Dates: Start 2005-08

PRIMARY OUTCOMES:
Peak increase in SCr
Incidence of contrast media-induced nephropathy from baseline up to day 3.

SECONDARY OUTCOMES:
SCr concentrations up to days 3 and 7
image quality
occurrence of adverse events and their severity and relationship with the contrast media.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Widlund, BSc RN, Study Director — GE Healthcare; Johnny Gibbs, Jr., B.S., CCRA, Study Director — 609-514-6809
Locations (1):
- Amersham Health S.A, Solna, Sweden

REFERENCES:
- [Derived] Laskey W, Aspelin P, Davidson C, Rudnick M, Aubry P, Kumar S, Gietzen F, Wiemer M; DXV405 Study Group. Nephrotoxicity of iodixanol versus iopamidol in patients with chronic kidney disease and diabetes mellitus undergoing coronary angiographic procedures. Am Heart J. 2009 Nov;158(5):822-828.e3. doi: 10.1016/j.ahj.2009.08.016. PMID 19853704